CLINICAL TRIAL: NCT00940394
Title: Evaluation of the Effects of Mutual Support and Psycho-educational Group Interventions for Family Caregivers of People With Schizophrenia
Brief Title: Effectiveness of Family Group Interventions for People With Schizophrenia
Acronym: MSG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Chien Wai-Tong, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 216020
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Schizophrenia
Keywords: mutual support group; psychoeducation group; family caregivers; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- standard care (Other): Families receive routine community and family mental health care services
  Interventions: Other: Standard care
- mutual support group (Experimental): bi-weekly, 12-session, family-led mutual support group
  Interventions: Behavioral: mutual support group
- psychoeducation group (Active Comparator): bi-weekly, 12-session, family psychoeducation group program
  Interventions: Behavioral: psychoeducation group

INTERVENTIONS:
Behavioral: mutual support group — bi-weekly, 12-session, family-led mutual support group
  Other Names: FMSG
  Arms: mutual support group
Behavioral: psychoeducation group — bi-weekly, 12-session, family psychoeducation group
  Other Names: FPGP
  Arms: psychoeducation group
Other: Standard care — Routine mental health care services provided by the outpatient clinic and related agencies for families of people with schizophrenia
  Other Names: Usual psychiatric care
  Arms: standard care

SUMMARY:
The mutual support group intervention would significantly improve the families' burden of care, functioning and social support, reduce the patients' severity of symptoms and re-hospitalizations, and reduce the demands for utilization of family services, when compared with the standard care group.

DETAILED DESCRIPTION:
Family interventions in schizophrenia have shown positive effects on patients but little attention has been paid to their effects on family members, particularly those in non-Western countries. This multi-site randomized controlled trial evaluated the effectiveness of a bi-weekly, 12-session, family-led mutual support group for Chinese caregivers of schizophrenia sufferers over 36 months, compared with a family psychoeducation group program and standard psychiatric care. It was conducted with 114 families of outpatients with schizophrenia in Hong Kong of whom 38 were assigned randomly to a mutual support group, a psychoeducation group, or standard care. Families' psychosocial health status and patients' symptom severity and length of re-hospitalizations at recruitment, one-month, 18-month, and 36-month post-intervention were compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* family caregivers lived with and cared for one family member diagnosed with schizophrenia according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV; American Psychiatric Association, 1994)
* family caregivers were at least 18 years of age and could understand and read the Chinese (Mandarin) language; and
* family caregivers were free from any mental illness themselves.

Exclusion Criteria:

* the patients with schizophrenia suffered no co-morbidity due to other mental illness during recruitment to the study
* family caregivers cared for more than one family member with mental or chronic physical illness; and/or
* family caregivers had been the primary carers for less than three months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2007-01; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
length of re-hospitalizations | at recruitment, six-month, 18-month and 36-month post-intervention

SECONDARY OUTCOMES:
families' perceived social support | at recruitment, six-month, 18-month and 36-month post-intervention
patients' symptom severity | at recruitment, six-month, 18-month and 36-month post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Chien Wai-Tong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- Hong Kong (2):
  - Li Ka Shing Specialty OPD, Shatin, NT
  - AHNH Psychiatric OPD, Taipo, NT

REFERENCES:
- [Result] Chien WT, Thompson DR, Norman I. Evaluation of a peer-led mutual support group for Chinese families of people with schizophrenia. Am J Community Psychol. 2008 Sep;42(1-2):122-34. doi: 10.1007/s10464-008-9178-8. PMID 18584319
- [Result] Chien WT, Thompson DR. An RCT with three-year follow-up of peer support groups for Chinese families of persons with schizophrenia. Psychiatr Serv. 2013 Oct;64(10):997-1005. doi: 10.1176/appi.ps.201200243. PMID 23820670
- [Result] Chien WT, Chan SW. The effectiveness of mutual support group intervention for Chinese families of people with schizophrenia: a randomised controlled trial with 24-month follow-up. Int J Nurs Stud. 2013 Oct;50(10):1326-40. doi: 10.1016/j.ijnurstu.2013.01.004. Epub 2013 Feb 19. PMID 23433723
- [Derived] Chien WT, Bressington D, Chan SWC. A Randomized Controlled Trial on Mutual Support Group Intervention for Families of People With Recent-Onset Psychosis: A Four-Year Follow-Up. Front Psychiatry. 2018 Dec 18;9:710. doi: 10.3389/fpsyt.2018.00710. eCollection 2018. PMID 30618880
- See also: Effectiveness of Psychoeducation and Mutual Support Group Program for Family Caregivers of Chinese People with Schizophrenia — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2582821/pdf/TONURSJ-2-28.pdf